CLINICAL TRIAL: NCT00993031
Title: Protease Inhibitors to Reduce Malaria Morbidity in HIV-Infected Pregnant Women
Acronym: PROMOTE-PIs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Diana Havlir, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H5741-34342; P01HD059454 (NIH); 2009-141 (Other: Makerere Univ Fac of Med Research and Ethics Committee); HS-670 (Other: Uganda National Council for Science and Tech); 592/ESR/NDA/DID-09/2009 (Other: Uganda National Drug Authority); H5741-34342 and 10-02958 (Other: UCSF Committee on Human Research)
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Malaria; HIV Infections
Keywords: HIV; Placental Malaria; Pregnancy; Uganda; Protease inhibitors; Trimethoprim-sulfamethoxazole; Treatment experienced
MeSH Terms: conditions — Malaria; HIV Infections | interventions — Lopinavir; lopinavir-ritonavir drug combination; efavirenz; Zidovudine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): ZDV 300mg/3TC 150mg/LPV 200mg/r 50mg
  Interventions: Drug: Lopinavir/ritonavir; Drug: Zidovudine; Drug: Lamivudine
- Group B (Active Comparator): ZDV 300mg/3TC 150mg/EFV 600mg
  Interventions: Drug: Efavirenz; Drug: Zidovudine; Drug: Lamivudine

INTERVENTIONS:
Drug: Lopinavir/ritonavir — LPV 200mg/r 50mg
  Other Names: Kaletra; Aluvia
  Arms: Group A
Drug: Efavirenz — 600mg
  Arms: Group B
Drug: Zidovudine — Zidovudine 300 mg
Drug: Lamivudine — Lamivudine 150 mg

SUMMARY:
This study is an open-label, single site, randomized controlled trial comparing protease inhibitor (PI)-based antiretroviral therapy (ART) to non-PI based ART for HIV-infected pregnant and breastfeeding women of all CD4 cell counts at high risk of malaria. The study is designed to test the hypothesis that pregnant women receiving a PI-based ART regimen will have lower risk of placental malaria compared to pregnant women receiving a non-PI based ART regimen. The primary study endpoint of the study is placental malaria. This study also enrolls the infants of these women at the time of delivery.

DETAILED DESCRIPTION:
The study site will be the Tororo district hospital campus situated in Eastern Uganda, an area of high malaria transmission. Using convenience sampling, we will enroll 500 HIV-infected pregnant women and their infants from the Tororo community. Eligible women between 12-28 weeks gestation will be randomized at enrollment to receive either a PI- based or an NNRTI-based ART regimen after stratification by gravidity (G1 versus G2+) and gestational age (<24 weeks versus ≥ 24 weeks at enrollment).

Treatment group A will receive Zidovudine 300mg + Lamivudine 150mg + Lopinavir/ritonavir 200mg/50mg. Treatment group B will receive Zidovudine 300mg + Lamivudine 150mg + Efavirenz 600mg.

At enrollment, all study participants will receive a long lasting ITN and, as available, a basic care package including a safe water vessel, multivitamins and condoms, as per current standard of care for HIV-infected pregnant women in Uganda, if they have not already received these interventions from the referral site. Two ITNs will be provided for each mother-infant pair. Participants will receive all routine and acute medical care at a designated study clinic open 7 days a week from 8 a.m. to 5 p.m. If medical care is needed after hours, participants will be instructed to come to Tororo District Hospital premises (where the study clinic is located) and request that the study physician on-call be contacted. They will be followed up from the time of enrollment during pregnancy and through the cessation of breastfeeding; seen monthly for routine assessments and laboratory evaluations. Following delivery, the infants of enrolled women will be followed until 6 weeks following the cessation of breastfeeding but not beyond 58 weeks of life. Study participants will be followed closely for adverse events potentially due to study drugs and for malaria and HIV treatment outcomes. During the follow-up period, all patients presenting to the clinic with a new episode of fever will undergo standard evaluation (history, physical examination and Giemsa-stained blood smear) for the diagnosis of malaria.

Women will receive the study treatment from the time of study entry and randomization (12-28 weeks gestation) until 1 week following the cessation of breastfeeding (but no longer than 1 year + 1 week postpartum). If a subject experiences a toxicity endpoint, ART will be changed to provide antiviral activity prior to delivery. Exclusive breastfeeding will be encouraged until 24 weeks postpartum which is the standard of care in Uganda. As per updated WHO guidelines, women will be encouraged to introduce food at 6 months of life and continue breastfeeding until 1 year of life. Women will be counseled to wean over the course of 1 month and continue antiretrovirals for at least 1 week following weaning. Furthermore, if an infant is found to be HIV-infected, Uganda MOH and WHO guidelines recommend the continuation of breastfeeding until 2 years of life and daily TS. All women will receive daily oral trimethoprim/sulfamethoxazole (TS) per Ugandan MOH guidelines.

Per Ugandan MOH guidelines, all newborns will receive nevirapine syrup (10mg/ml) starting within 12 hours after birth for 6 weeks, daily oral TS from 6 weeks of life until 6 weeks following the cessation of breastfeeding, and their mothers will be instructed on ITN use for their infants.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 16 years (if <18 years old, living independently from parents)
2. Documentation of HIV status must come from two assays. Assays include DNA PCR, HIV RNA, Western blot, or rapid HIV antibody test
3. Confirmed pregnancy by positive serum or urine pregnancy test or ultrasound
4. Estimated gestational age between 12 and 28 weeks (based on first day of last menstrual period with physical exam confirmation and ultrasound confirmation) at time of enrollment
5. Residency within 30 km of the study site
6. Willing to provide informed consent

Exclusion Criteria:

1. Current or prior use of HAART
2. Exposure to single-dose NVP (alone or with zidovudine or zidovudine/lamivudine or other abbreviated monotherapy or dual therapy for PMTCT) less than 24 months prior to enrollment
3. Prior dose-limited toxicity to TS within 14 days of study enrollment
4. Receipt of any contraindicated medications within 14 days of study enrollment (See Appendix III.)
5. Active tuberculosis or other WHO Stage 4 diseases
6. Screening laboratory values:

   1. Hemoglobin: <7.5 g/dL (Note: Women found to have a hemoglobin <7.5 at screening may receive iron and folic acid and/or a blood transfusion at the physician's discretion. If a repeat hemoglobin is ≥7.5 g/dL, the woman may be considered for study inclusion.)
   2. Absolute neutrophil count (ANC): <750/mm3
   3. Platelet count: <50,000/mm3
   4. ALT: >225 U/L (>5.0x ULN)
   5. AST: >225 U/L (>5.0x ULN)
   6. Bilirubin (total): > 2.5x ULN
   7. Creatinine: > 1.8x ULN
7. Known cardiac conduction abnormalities or structural heart defect

NOTE: A woman will be excluded from study participation during the current pregnancy if she goes into labor, experiences ruptured membranes or develops active tuberculosis or a WHO stage 4 condition following study enrollment but prior to study drug initiation.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2009-12-15 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Principal Investigator — University of California, San Francisco; Deborah Cohan, MD, MPH, Study Chair — University of California, San Francisco; Moses R Kamya, MBChB, MMed, PhD, Principal Investigator — Makerere University; Pius Okong, MMed, PhD, Study Chair — Ugandan Ministry of Health; Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Tororo District Hospital, Tororo, Uganda

REFERENCES:
- [Background] Nsanzabana C, Rosenthal PJ. In vitro activity of antiretroviral drugs against Plasmodium falciparum. Antimicrob Agents Chemother. 2011 Nov;55(11):5073-7. doi: 10.1128/AAC.05130-11. Epub 2011 Aug 29. PMID 21876053
- [Background] Ochong E, Tumwebaze PK, Byaruhanga O, Greenhouse B, Rosenthal PJ. Fitness Consequences of Plasmodium falciparum pfmdr1 Polymorphisms Inferred from Ex Vivo Culture of Ugandan Parasites. Antimicrob Agents Chemother. 2013 Sep;57(9):4245-4251. doi: 10.1128/AAC.00161-13. Epub 2013 Jun 24. PMID 23796921
- [Result] Young S, Murray K, Mwesigwa J, Natureeba P, Osterbauer B, Achan J, Arinaitwe E, Clark T, Ades V, Plenty A, Charlebois E, Ruel T, Kamya M, Havlir D, Cohan D. Maternal nutritional status predicts adverse birth outcomes among HIV-infected rural Ugandan women receiving combination antiretroviral therapy. PLoS One. 2012;7(8):e41934. doi: 10.1371/journal.pone.0041934. Epub 2012 Aug 7. PMID 22879899
- [Result] Cohan D, Mwesigwa J, Natureeba P, Aliba Luwedde F, Ades V, Plenty A, Kakuru A, Achan J, Clark T, Osterbauer B, Kamya M, Havlir D. WHO option B+: early experience of antiretroviral therapy sequencing after cessation of breastfeeding and risk of dermatologic toxicity. J Acquir Immune Defic Syndr. 2013 Mar 1;62(3):e101-3. doi: 10.1097/QAI.0b013e31828011ca. No abstract available. PMID 23924639
- [Result] Ades V, Mwesigwa J, Natureeba P, Clark TD, Plenty A, Charlebois E, Achan J, Kamya MR, Havlir DV, Cohan D, Ruel TD. Neonatal mortality in HIV-exposed infants born to women receiving combination antiretroviral therapy in Rural Uganda. J Trop Pediatr. 2013 Dec;59(6):441-6. doi: 10.1093/tropej/fmt044. Epub 2013 Jun 13. PMID 23764539
- [Result] Bartelink IH, Savic RM, Mwesigwa J, Achan J, Clark T, Plenty A, Charlebois E, Kamya M, Young SL, Gandhi M, Havlir D, Cohan D, Aweeka F. Pharmacokinetics of lopinavir/ritonavir and efavirenz in food insecure HIV-infected pregnant and breastfeeding women in Tororo, Uganda. J Clin Pharmacol. 2014 Feb;54(2):121-32. doi: 10.1002/jcph.167. Epub 2013 Sep 21. PMID 24038035
- [Result] Gandhi M, Mwesigwa J, Aweeka F, Plenty A, Charlebois E, Ruel TD, Huang Y, Clark T, Ades V, Natureeba P, Luwedde FA, Achan J, Kamya MR, Havlir DV, Cohan D; Prevention of Malaria and HIV disease in Tororo (PROMOTE) study. Hair and plasma data show that lopinavir, ritonavir, and efavirenz all transfer from mother to infant in utero, but only efavirenz transfers via breastfeeding. J Acquir Immune Defic Syndr. 2013 Aug 15;63(5):578-84. doi: 10.1097/QAI.0b013e31829c48ad. PMID 24135775
- [Result] Young SL, Plenty AH, Luwedde FA, Natamba BK, Natureeba P, Achan J, Mwesigwa J, Ruel TD, Ades V, Osterbauer B, Clark TD, Dorsey G, Charlebois ED, Kamya M, Havlir DV, Cohan DL. Household food insecurity, maternal nutritional status, and infant feeding practices among HIV-infected Ugandan women receiving combination antiretroviral therapy. Matern Child Health J. 2014 Nov;18(9):2044-53. doi: 10.1007/s10995-014-1450-y. PMID 24585398
- [Result] Natureeba P, Ades V, Luwedde F, Mwesigwa J, Plenty A, Okong P, Charlebois ED, Clark TD, Nzarubara B, Havlir DV, Achan J, Kamya MR, Cohan D, Dorsey G. Lopinavir/ritonavir-based antiretroviral treatment (ART) versus efavirenz-based ART for the prevention of malaria among HIV-infected pregnant women. J Infect Dis. 2014 Dec 15;210(12):1938-45. doi: 10.1093/infdis/jiu346. Epub 2014 Jun 23. PMID 24958908
- [Result] Koss CA, Natureeba P, Plenty A, Luwedde F, Mwesigwa J, Ades V, Charlebois ED, Clark TD, Achan J, Ruel T, Nzarubara B, Kamya MR, Havlir DV, Cohan D. Risk factors for preterm birth among HIV-infected pregnant Ugandan women randomized to lopinavir/ritonavir- or efavirenz-based antiretroviral therapy. J Acquir Immune Defic Syndr. 2014 Oct 1;67(2):128-35. doi: 10.1097/QAI.0000000000000281. PMID 25072616
- [Result] Cohan D, Natureeba P, Koss CA, Plenty A, Luwedde F, Mwesigwa J, Ades V, Charlebois ED, Gandhi M, Clark TD, Nzarubara B, Achan J, Ruel T, Kamya MR, Havlir DV. Efficacy and safety of lopinavir/ritonavir versus efavirenz-based antiretroviral therapy in HIV-infected pregnant Ugandan women. AIDS. 2015 Jan 14;29(2):183-91. doi: 10.1097/QAD.0000000000000531. PMID 25426808
- [Result] Young S, Natamba B, Luwedde F, Nyafwono D, Okia B, Osterbauer B, Natureeba P, Johnson L, Michel C, Zheng A, Robine M, Achan J, Charlebois E, Cohan D, Havlir D. "I Have Remained Strong Because of That Food": Acceptability and Use of Lipid-Based Nutrient Supplements Among Pregnant HIV-Infected Ugandan Women Receiving Combination Antiretroviral Therapy. AIDS Behav. 2015 Aug;19(8):1535-47. doi: 10.1007/s10461-014-0947-0. PMID 25416075
- [Result] Koss CA, Natureeba P, Mwesigwa J, Cohan D, Nzarubara B, Bacchetti P, Horng H, Clark TD, Plenty A, Ruel TD, Achan J, Charlebois ED, Kamya MR, Havlir DV, Gandhi M. Hair concentrations of antiretrovirals predict viral suppression in HIV-infected pregnant and breastfeeding Ugandan women. AIDS. 2015 Apr 24;29(7):825-30. doi: 10.1097/QAD.0000000000000619. PMID 25985404
- [Result] Koss CA, Natureeba P, Nyafwono D, Plenty A, Mwesigwa J, Nzarubara B, Clark TD, Ruel TD, Achan J, Charlebois ED, Cohan D, Kamya MR, Havlir DV, Young SL. Brief Report: Food Insufficiency Is Associated With Lack of Sustained Viral Suppression Among HIV-Infected Pregnant and Breastfeeding Ugandan Women. J Acquir Immune Defic Syndr. 2016 Mar 1;71(3):310-5. doi: 10.1097/QAI.0000000000000860. PMID 26397935
- [Result] Marquez C, Chamie G, Achan J, Luetkemeyer AF, Kyohere M, Okiring J, Dorsey G, Kamya MR, Charlebois ED, Havlir DV. Tuberculosis Infection in Early Childhood and the Association with HIV-exposure in HIV-uninfected Children in Rural Uganda. Pediatr Infect Dis J. 2016 May;35(5):524-9. doi: 10.1097/INF.0000000000001062. PMID 26771662
- [Result] Parikh S, Kajubi R, Huang L, Ssebuliba J, Kiconco S, Gao Q, Li F, Were M, Kakuru A, Achan J, Mwebaza N, Aweeka FT. Antiretroviral Choice for HIV Impacts Antimalarial Exposure and Treatment Outcomes in Ugandan Children. Clin Infect Dis. 2016 Aug 1;63(3):414-22. doi: 10.1093/cid/ciw291. Epub 2016 May 3. PMID 27143666
- [Result] Koss CA, Natureeba P, Kwarisiima D, Ogena M, Clark TD, Olwoch P, Cohan D, Okiring J, Charlebois ED, Kamya MR, Havlir DV. Viral Suppression and Retention in Care up to 5 Years After Initiation of Lifelong ART During Pregnancy (Option B+) in Rural Uganda. J Acquir Immune Defic Syndr. 2017 Mar 1;74(3):279-284. doi: 10.1097/QAI.0000000000001228. PMID 27828878
- [Result] Kakuru A, Natureeba P, Muhindo MK, Clark TD, Havlir DV, Cohan D, Dorsey G, Kamya MR, Ruel T. Malaria burden in a birth cohort of HIV-exposed uninfected Ugandan infants living in a high malaria transmission setting. Malar J. 2016 Oct 18;15(1):500. doi: 10.1186/s12936-016-1568-z. PMID 27756308
- [Derived] Finkelstein JL, Herman HS, Plenty A, Mehta S, Natureeba P, Clark TD, Kamya MR, Ruel T, Charlebois ED, Cohan D, Havlir D, Young SL. Anemia and Micronutrient Status during Pregnancy, and Their Associations with Obstetric and Infant Outcomes among HIV-Infected Ugandan Women Receiving Antiretroviral Therapy. Curr Dev Nutr. 2020 Apr 25;4(5):nzaa075. doi: 10.1093/cdn/nzaa075. eCollection 2020 May. PMID 32440638
- [Derived] McDonald CR, Conroy AL, Gamble JL, Papp E, Hawkes M, Olwoch P, Natureeba P, Kamya M, Silverman M, Cohan D, Koss CA, Dorsey G, Kain KC, Serghides L. Estradiol Levels Are Altered in Human Immunodeficiency Virus-Infected Pregnant Women Randomized to Efavirenz-Versus Lopinavir/Ritonavir-Based Antiretroviral Therapy. Clin Infect Dis. 2018 Jan 18;66(3):428-436. doi: 10.1093/cid/cix772. PMID 29136115

RESULTS

PARTICIPANT FLOW:
Groups:
- Without Protease Inhibitor: ZDV 300mg/3TC 150mg/EFV 600mg
  Efavirenz: 600mg
  Zidovudine: Zidovudine 300 mg
  Lamivudine: Lamivudine 150 mg
- With Protease Inhibitor: ZDV 300mg/3TC 150mg/LPV 200mg/r 50mg
  Lopinavir/ritonavir: LPV 200mg/r 50mg
  Zidovudine: Zidovudine 300 mg
  Lamivudine: Lamivudine 150 mg
Period: Overall Study
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor
Started | 195 | 194
Delivered | 187 | 190
Completed | 173 | 175
Not Completed | 22 | 19
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 19 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor | Total
Number analyzed (Participants) | 195 | 194 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.4) | 29.0 (5.4) | 29.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 194 | 389
  Male | 0 | 0 | 0
Gestational Age, wk [Mean (Standard Deviation); unit: weeks] | 21.1 (4.1) | 21.2 (4.3) | 21.1 (5.9)
Previous Preganancies [Number; unit: participants]
  0 | 16 | 8 | 24
  1 | 20 | 25 | 45
  ≥2 | 159 | 161 | 320
Bed Net Ownership [Number; unit: participants]
  None | 85 | 85 | 170
  Untreated | 28 | 33 | 61
  ITN | 77 | 70 | 147
  Yes; unknown treatment status | 5 | 5 | 10
  Unknown | 0 | 1 | 1
Receiving TMP-SMX prophylaxis at enrollment [Number; unit: participants] — Trimethoprim/sulfamethoxazole (TMP-SMX) is an antibiotic used to treat a variety of bacterial infections. It consists of one part trimethoprim to five parts sulfamethoxazole.
  participants | 125 | 124 | 249
Hemoglobin level, g/dL [Mean (Standard Deviation); unit: g/dL] | 10.9 (1.3) | 11.0 (1.2) | 10.9 (1.8)
CD4+ T-cell count [Median (Inter-Quartile Range); unit: cells/mm3] | 374 [270 to 485] | 368 [282 to 506] | 370.5 [274 to 494]
HIV RNA load [Median (Inter-Quartile Range); unit: log10 copies/mL] | 4.3 [3.5 to 4.8] | 4.1 [3.3 to 4.7] | 4.1 [3.4 to 4.8]
WHO stage HIV disease [Number; unit: participants] — Stage 1=Asymptomatic; Stage 2= Moderate unexplained weight loss, Recurrent respiratory infections, Herpes zoster, Angular cheilitis, Recurrent oral ulceration, Papular pruritic eruptions, Seborrheic dermatitis, Fungal nail infections; Stage 3=Unexplained severe weight loss, Unexplained chronic diarrhea for >1 month, Unexplained persistent fever for >1 month, Persistent oral candidiasis, Oral hairy leukoplakia, Pulmonary tuberculosis, Severe presumed bacterial infections, Acute necrotizing ulcerative stomatitis, gingivitis, or periodontitis; Unexplained anemia; Stage 4 =HIV wasting syndrome,etc
  participants
    1 | 181 | 189 | 370
    2 | 13 | 5 | 18
    3 | 1 | 0 | 1
    4 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Malaria Defined as Positive Placental Blood Smear
Description: Number of participants with positive placental blood smear for malaria
Time Frame: Delivery
Population: Placental blood smear
Measure: Number; unit: participants
Arm/Group | With Protease Inhibitor | Without Protease Inhibitor
Number analyzed (Participants) | 158 | 158
participants | 5 | 6
Statistical Analysis 1: Comparison: With Protease Inhibitor vs Without Protease Inhibitor; Test type: Superiority or Other; p = .76, Chi-squared; Risk Ratio (RR) = 0.83, 95% CI 2-sided [.26 to 2.67]

2. Primary Outcome: Prevalence of Malaria Defined as Positive Placental Blood PCR
Description: Number of participants with positive placental blood PCR for malaria
Time Frame: Delivery
Population: Placental blood PCR
Measure: Number; unit: participants
Arm/Group | With Protease Inhibitor | Without Protease Inhibitor
Number analyzed (Participants) | 157 | 155
participants | 6 | 7
Statistical Analysis 1: Comparison: With Protease Inhibitor vs Without Protease Inhibitor; Test type: Superiority or Other; p = .76, Chi-squared; Risk Ratio (RR) = .85, 95% CI 2-sided [.29 to 2.46]

3. Secondary Outcome: Placental Malaria Defined as Positive Placental RDT
Description: Number of participants with positive placental RDT for malaria. Malaria rapid diagnostic tests (RDTs) assist in the diagnosis of malaria by detecting evidence of malaria parasites (antigens) in human blood. RDTs permit a reliable detection of malaria infections particularly in remote areas with limited access to good quality microscopy services.
Time Frame: Delivery
Population: Some participants did not have a placental specimen taken at delivery in the hospital (e.g. deliveries that occurred at home, missed by staff error, etc)
Measure: Number; unit: participants
Arm/Group | With Protease Inhibitor | Without Protease Inhibitor
Number analyzed (Participants) | 157 | 155
participants | 6 | 7
Statistical Analysis 1: Comparison: With Protease Inhibitor vs Without Protease Inhibitor; Test type: Superiority or Other; p = .45, Chi-squared; Risk Ratio (RR) = .75, 95% CI 2-sided [.36 to 1.59]

4. Secondary Outcome: Maternal Malaria Defined as the Number of Treatments for New Episodes of Malaria Per Time at Risk During Pregnancy
Time Frame: Number of treatments given for clinical malaria based on postive blood smear from time from randomization until 24 months after delivery or cessation of breastfeeding
Measure: Number; unit: treatments
Arm/Group | With Protease Inhibitor | Without Protease Inhibitor
Number analyzed (Participants) | 194 | 195
treatments | 17 | 17

5. Secondary Outcome: Prevalence of Composite Clinical Outcome Defined by LBW, Stillbirth(Intrauterine Fetal Demise >20wks GA), Late Spontaneous Abortion(Miscarriage 12-20wks GA), Preterm Delivery(<37wks Gestation), Neonatal Death(Death of Liveborn Infant Within First 28days)
Description: Percent of evaluated participants with composite clinical outcome defined by LBW, stillbirth (intrauterine fetal demise >20wks GA), late spontaneous abortion(miscarriage 12-20wks GA), preterm delivery(<37wks gestation), neonatal death(death of live-born infant within first 28 days)
Time Frame: Time from randomization until 24 months postpartum or cessation of breastfeeding
Measure: Number; unit: % of evaluated participants with outcome
Arm/Group | With Protease Inhibitor | Without Protease Inhibitor
Number analyzed (Participants) | 186 | 180
% of evaluated participants with outcome | 33.9 | 27.8
Statistical Analysis 1: Comparison: With Protease Inhibitor vs Without Protease Inhibitor; Test type: Superiority or Other; p = .21, Chi-squared; Risk Ratio (RR) = 1.22, 95% CI 2-sided [.89 to 1.66]

6. Secondary Outcome: Placental Malaria Defined Placental Histopathologic Analysis
Description: Number of participants with positive placental histopathology slide for malaria
Time Frame: Delivery
Measure: Number; unit: participants
Arm/Group | With Protease Inhibitor | Without Protease Inhibitor
Number analyzed (Participants) | 162 | 165
participants | 62 | 47
Statistical Analysis 1: Comparison: With Protease Inhibitor vs Without Protease Inhibitor; Test type: Superiority or Other; p = .06, Chi-squared; Risk Ratio (RR) = 1.34, 95% CI 2-sided [.98 to 1.83]

7. Secondary Outcome: Maternal Malaria Defined as the Number of Treatments for New Episodes of Malaria Per Time at Risk After Pregnancy
Time Frame: Number of treatments given for clinical malaria based on postive blood smear from time from delivery until 24 months after delivery or cessation of breastfeeding
Measure: Number; unit: treatments
Arm/Group | Group A | Group B
Number analyzed (Participants) | 190 | 187
treatments | 21 | 13

8. Secondary Outcome: Number of Participants With Severe Maternal Anemia Defined by Hemoglobin < 8g/dl at Any Point During the Trial in Each Treatment Group
Description: Proportion of women with severe maternal Anemia (hemoglobin < 8g/dl by hemacue or CBC) at any point during the trial in Each Treatment Group
Time Frame: Time from randomization until one year follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor
Number analyzed (Participants) | 195 | 194
Participants | 11 | 11

9. Secondary Outcome: Incidence of Pre-eclampsia Defined by Hypertension > 140/90 on Two Occasions Measured > 6 Hours Apart With ≥1+ Proteinuria on Clean Catch Urine Dipstick
Description: Pre-eclampsia Defined by Hypertension > 140/90 on Two Occasions Measured > 6 Hours Apart With ≥1+ Proteinuria on Clean Catch Urine Dipstick
Time Frame: Time from randomization until delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor
Number analyzed (Participants) | 187 | 190
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Maternal HIV RNA Suppression of <400 Copies/mL
Description: Virologic suppression was defined as plasma HIV-1 RNA 400 copies/ml or less based on the lower limit of detection of the available test.
Time Frame: Time from randomization until delivery, an average of 20 weeks
Population: Note: The above numbers differ from the numbers of participants who delivered according to the Patient Flow Overview (187 and 190, respectively) due to the inability to measure HIV RNA a small number of women at delivery, for technical or logistical reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor
Number analyzed (Participants) | 170 | 178
Participants | 166 | 153

11. Secondary Outcome: Change in Maternal CD4 Cell Counts
Description: CD4 cell count recovery efavirenz at delivery
Time Frame: Time of randomization to delivery, an average of 20 weeks
Measure: Median (Standard Deviation); unit: CD4 cell count
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor
Number analyzed (Participants) | 195 | 194
CD4 cell count | -7 (.002) | 57 (.002)

12. Secondary Outcome: Number of Participants With Maternal to Child Transmission of HIV, Measured by Infant HIV DNA PCR
Description: HIV tested by DNA PCR
Time Frame: Delivery to 48 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor
Number analyzed (Participants) | 195 | 194
Participants | 0 | 2

13. Secondary Outcome: ART Levels in Hair Samples at Delivery
Description: antiretroviral hair concentrations (per doubling)
Time Frame: delivery
Population: Note: The above numbers differ from the numbers of participants who delivered according to the Patient Flow Overview (187 and 190, respectively) due to the fact that a small number participants chose to decline this optional measurement.
Measure: Mean (Full Range); unit: antiretroviral hair concentration(ng/mg)
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor
Number analyzed (Participants) | 162 | 163
antiretroviral hair concentration(ng/mg) | 5.7 [0.05 to 36.7] | 6.6 [0.05 to 47.2]

14. Secondary Outcome: Number of Participants With Grade 3 or 4 Toxicity in the Two Treatment Groups in Women
Time Frame: Randomization to one month postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Without Protease Inhibitor | With Protease Inhibitor
Number analyzed (Participants) | 195 | 194
Participants | 12 | 8

ADVERSE EVENTS:
Time Frame: Gestational age between 12 and 28 weeks at time of enrollment up to at least 1 year of follow up after delivery or until study termination.
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 28/194 | 32/195
Other Adverse Events (participants affected / at risk) | 140/194 | 137/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=194) | Group B (N=195)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Complicated malaria (Infections and infestations) | 0 (0) | 1 (1)
Death, natural causes (General disorders) | 2 (2) | 0 (0)
Deep venous Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Abruptio-placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Antepartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Severe anemia (Hepatobiliary disorders) | 7 (7) | 5 (5)
Neutropenia (Hepatobiliary disorders) | 9 (9) | 5 (5)
Thrombocytopenia (Hepatobiliary disorders) | 2 (2) | 3 (3)
Abdominal pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Intra-uterine fetal death (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 5 (5)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Preterm contractions (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3)
Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pyelonephritis (Hepatobiliary disorders) | 3 (3) | 1 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=194) | Group B (N=195)
Abdominal pain (General disorders) | 63 (84) | 46 (64)
Altered mental status (Psychiatric disorders) | 0 (0) | 1 (1)
Anemia (Hepatobiliary disorders) | 18 (34) | 24 (33)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 8 (14)
Chills (General disorders) | 8 (8) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (33) | 19 (36)
Deep vein thrombosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 6 (10)
Dizziness/Lightheadedness (General disorders) | 2 (2) | 4 (4)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Dysphagia/odynophagia (General disorders) | 1 (1) | 2 (2)
Dyspnea/respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 5 (16)
Elevated ALT (Renal and urinary disorders) | 3 (4) | 6 (7)
Elevated AST (Renal and urinary disorders) | 4 (4) | 0 (0)
Elevated bilirubin (Renal and urinary disorders) | 0 (0) | 1 (1)
Fatigue/malaise (General disorders) | 33 (39) | 26 (37)
Headache (General disorders) | 15 (19) | 11 (13)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Nausea (General disorders) | 5 (5) | 3 (3)
Neurosensory alteration (Psychiatric disorders) | 2 (2) | 2 (6)
Neutropenia (Blood and lymphatic system disorders) | 58 (100) | 62 (130)
Oral sores (General disorders) | 0 (0) | 1 (7)
Pain, general (General disorders) | 15 (17) | 16 (21)
Pallor (Blood and lymphatic system disorders) | 4 (5) | 1 (5)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pre-term premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 5 (7) | 4 (5)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 3 (3)
Rash (non-infectious) (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Reduced WBC count (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
Serum glucose, low (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Temperature, elevated (General disorders) | 10 (11) | 7 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (23) | 11 (24)
Unintentional weight loss (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Urine Protein (Renal and urinary disorders) | 41 (47) | 25 (33)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 0 (0)

LIMITATIONS AND CAVEATS:
A semi-immune population of adults at relatively low risk for malaria; a high rate of TMP-SMX prophylaxis ; A lower than expected incidence of malaria, resulting in the possibility that the study was underpowered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No